CLINICAL TRIAL: NCT05897827
Title: Providing LGBTQ+ Adolescents With Nurturance, Trustworthiness, and Safety (PLANTS): Pilot Cluster-Randomized Controlled Trial
Brief Title: PLANTS Pilot Trial
Acronym: PLANTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Robert Coulter, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY23040142; K01AA027564 (NIH)
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Drinking; Social Acceptance; Depressive Symptoms; Bullying
Keywords: Sexual and gender minority youth
MeSH Terms: conditions — Alcohol Drinking; Depression; Bullying; Coitus | interventions — Safety

STUDY DESIGN:
Intervention Model Description: This is a two-armed cluster-randomized controlled pilot trial of the PLANTS intervention versus an active control group, the EMAILS intervention. The investigators will randomize schools in an equal 1:1 ratio, stratified by large versus small schools, into intervention or active control conditions. The investigators will use block randomization with block sizes of 2, which will be stratified by large schools versus not, where large is ≥1000 students. The investigators use block size of 2 because there are only 4 schools in this pilot trial.
Masking Description: This is an unblinded study. This is an educational intervention that cannot be blinded because study participants will be able to tell which condition they are in based on the content they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLANTS (Experimental): Schools will receive the online-delivered PLANTS intervention, which includes 3 asynchronous training modules and 3 synchronous group events.
  Interventions: Behavioral: PLANTS
- EMAILS (Active Comparator): Comparison schools will receive emails with publicly available resources for supporting LGBTQ+ students as a control intervention.
  Interventions: Behavioral: EMAILS

INTERVENTIONS:
Behavioral: PLANTS — PLANTS intervention is an online-delivered training program, including asynchronous and synchronous activities. This intervention was informed by the Information-Motivation-Behavior theory to target skills, self-efficacy, knowledge, and outcome expectations. There are 3 asynchronous online modules that cover a variety of topics including lessons on LGBTQ+ terminology, names and pronouns, resources, antibullying, gender neutral bathrooms, student confidentiality, active empathic listening, and school policies. Module include recorded presentations, student testimonials, activities, and downloadable resources for future reference. Every month, 7-9 lessons are opened. There are 2 synchronous group events delivered via Zoom and are 1.5 hours each.
  Other Names: Providing LGBTQ+ Adolescents with Nurturance, Trustworthiness, and Safety
  Arms: PLANTS
Behavioral: EMAILS — The active control arm is an email-based intervention, EMAILS, in which existing public resources for supporting, affirming, and protecting LGBTQ+ students are emailed to participants.
  Other Names: E-learning to Maximize Academic Inclusion of LGBTQ+ Students
  Arms: EMAILS

SUMMARY:
This pilot cluster-randomized controlled trial will evaluate the PLANTS (Providing LGBTQ+ Adolescents with Nurturance, Trustworthiness, and Safety) course among high school staff. The primary hypotheses are that the PLANTS course will have high acceptability, usability, appropriateness, and feasibility as reported by high school staff.

DETAILED DESCRIPTION:
The intervention being studied, PLANTS, is an online-delivered training program, including asynchronous and synchronous activities targeting high school staff. This intervention is informed by the Information-Motivation-Behavior theory to target high school staffs' skills, self-efficacy, knowledge, and outcome expectations. Members of the study population as well as collaborators invested in Sexual and Gender Minority Youth (SGMY) well-being provided valuable feedback on PLANTS throughout its development. Comparison schools will receive the email-based control intervention, E-learning to Maximize Academic Inclusion of LGBTQ+ Students (EMAILS). Staff will receive periodic emails with publicly available resources on similar topics to those of PLANTS.

Regarding the intervention's targeted behavioral outcomes, upon completion of the PLANTS program, high school staff will: provide interpersonal support and affirmation to SGMY; provide educational resources that are inclusive of SGMY; provide safe spaces for SGMY; promote acceptance of SGMY among cisgender heterosexual youth; prevent and reduce bullying, cyberbullying, and harassment of SGMY; evaluate and advocate for SGMY inclusivity and protections in school policies; and maintain the confidentiality of SGMY. By having high school staff achieve these behavioral outcomes, the investigators hypothesize that SGMY will experience less risk factors (e.g., bullying victimization) and more protective factors (e.g., school-based adult support), which will in turn reduce SGMY's substance use and mental health problems.

The primary aim of this clinical trial is to rigorously test the acceptability, usability, appropriateness, and feasibility of the PLANTS intervention using a 2-armed cluster-randomized controlled trial. The investigators will also examine the efficacy of intervention in improving high school staff outcomes as well as implementation and safety outcomes related to the intervention and trial. Results from this pilot trial will provide necessary information to conduct a fully powered trial of the efficacy of PLANTS for reducing the ultimate health outcome of SGMY alcohol use.

ELIGIBILITY:
Inclusion Criteria:

* Currently employed by an enrolled school in the MetroWest Region of Boston, Massachusetts
* Age 18 years old or older
* Consents to participate

Exclusion Criteria:

• Does not interact with high school students at work

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Coulter, PhD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coulter RW, Mahal IK, Lin CA, Schneider SK, Mathias AS, Baral K, Miller E, Abebe KZ. Providing Lesbian, Gay, Bisexual, Transgender, Nonbinary, and Queer Adolescents With Nurturance, Trustworthiness, and Safety: Protocol for Pilot Cluster Randomized Controlled Trial Design. JMIR Res Protoc. 2024 Mar 19;13:e55210. doi: 10.2196/55210. PMID 38502156

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this pilot study, fewer school staff joined this study than anticipated.
Units Other Than Participants: Schools
Period: Overall Study
Arm/Group | PLANTS | EMAILS
Started | 69; 2 Schools | 30; 1 Schools
Completed Baseline Survey | 67; 2 Schools | 28; 1 Schools
Completed Follow-up Survey | 35; 2 Schools | 15; 1 Schools
Invited to Follow-up Interview | 22; 2 Schools | 10; 1 Schools
Completed Follow-up Interview | 13; 2 Schools | 6; 1 Schools
Completed | 35; 2 Schools | 15; 1 Schools
Not Completed | 34; 0 Schools | 15; 0 Schools
Not completed — Lost to Follow-up | 33 | 14
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Our baseline analysis population is the 67 participants from PLANTS and 28 participants from EMAILS who completed the baseline survey. It excludes the two participants (one from each arm) who never started baseline and the two participants (one from each arm) who did not complete the baseline survey.
Groups:
- Total: Total of all reporting groups
Arm/Group | PLANTS | EMAILS | Total
Number analyzed (Participants) | 67 | 28 | 95
Age, Continuous [Mean (Full Range); unit: years] | 44.04 [25 to 65] | 44.90 [23 to 65] | 44.30 [23 to 65]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Cisgender woman | 51 | 19 | 70
  Cisgender man | 15 | 9 | 24
  Nonbinary | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
  Hispanic | 1 | 1 | 2
  White | 65 | 25 | 90
  Unknown | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 67 | 28 | 95
Years Worked at School [Mean (Full Range); unit: years] | 16.34 [1 to 31] | 17.44 [3 to 27] | 16.65 [1 to 31]
Role in School [Count of Participants; unit: Participants]
  Teacher | 45 | 19 | 64
  Special education teacher | 5 | 2 | 7
  Administrator | 2 | 3 | 5
  Counselor or psychologist | 4 | 1 | 5
  Paraprofessional, teacher assistant, or instructional aide | 2 | 1 | 3
  Other certified staff | 3 | 1 | 4
  Multiple roles | 5 | 0 | 5
  Unknown | 1 | 1 | 2
Education Completed [Count of Participants; unit: Participants]
  Some college | 1 | 1 | 2
  Bachelor's degree | 6 | 0 | 6
  Master's degree | 55 | 25 | 80
  Professional degree beyond bachelor's degree | 2 | 1 | 3
  Doctorate degree | 3 | 1 | 4
Sexual Identity [Count of Participants; unit: Participants]
  Heterosexual (straight) | 58 | 22 | 80
  Gay or lesbian | 7 | 3 | 10
  Bisexual | 2 | 1 | 3
  Queer | 0 | 2 | 2
Current Religion [Count of Participants; unit: Participants]
  None | 44 | 16 | 60
  Catholicism | 14 | 5 | 19
  Judaism | 2 | 2 | 4
  Protestantism | 4 | 1 | 5
  Something Else | 1 | 2 | 3
  Multiple Religions | 1 | 1 | 2
  Unknown | 1 | 1 | 2
Childhood Religion [Count of Participants; unit: Participants]
  None | 9 | 5 | 14
  Catholicism | 41 | 15 | 56
  Judaism | 2 | 2 | 4
  Protestantism | 9 | 4 | 13
  Something else | 2 | 1 | 3
  Multiple religions | 2 | 0 | 2
  Unknown | 2 | 1 | 3
Religious Attendance [Mean (Standard Deviation); unit: units on a scale] — Duke University Religious Index (DUREL)
  Analyzed as the mean response to the item "How often do you attend religious meetings (e.g. church)?" where 1 means "Never" and 6 means "More than once/week".
  units on a scale | 2.16 (1.16) | 1.96 (1.07) | 2.11 (1.13)
Religious Activity [Mean (Standard Deviation); unit: units on a scale] — Duke University Religious Index (DUREL)
  Analyzed as the mean response to the item "How often do you spend time in private religious activities, such as prayer, meditation or Bible study?" where 1 means "Rarely or never" and 6 means "More than once a day".
  units on a scale | 1.90 (1.40) | 1.79 (1.34) | 1.86 (1.38)
Intrinsic Religiosity [Mean (Standard Deviation); unit: units on a scale] — Duke University Religion Index (DUREL)
  Calculated as the mean response across 3 items (ex. "In my life, I experience the presence of the Divine (i.e., God)"), each assessed from 1-5, where 1 means "Definitely not true" and 5 means "Definitely true". Higher values indicate more intrinsic religiosity.
  .
  units on a scale | 2.26 (1.12) | 1.96 (1.04) | 2.18 (1.10)
Social Desirability [Mean (Standard Deviation); unit: units on a scale] — Marlowe-Crowne Social Desirability Scale (13-item)
  Each participant receives a score from 0-13, where 1 point is added for a "True" or a "False", depending on the item. An example item is "No matter who I'm talking to, I'm always a good listener." A higher score indicates a tendency towards socially desirable responses.
  units on a scale | 4.71 (0.33) | 5.27 (0.50) | 4.88 (0.27)
Previous Training about LGBTQ+ Issues [Count of Participants; unit: Participants]
  Yes | 28 | 14 | 42
  No or not sure | 39 | 14 | 53
Previous Online Training about LGBTQ+ Issues [Count of Participants; unit: Participants]
  Yes | 3 | 7 | 10
  No or not sure | 64 | 21 | 85

OUTCOME MEASURES:

1. Primary Outcome: Mean Value of Acceptability of Intervention Measure
Description: At follow-up, participants will complete the four-question Acceptability of Intervention Measure (AIM) about PLANTS. Each question uses a five-point Likert scale for responses, coded with a value from 1 (Completely disagree) to 5 (Completely agree) and averaged to produce the mean acceptability value. The minimum possible mean value is 1 and the maximum mean value is 5. The higher the computed mean value, the more acceptable the intervention.
Time Frame: Approximately 4 months after intervention deployment
Population: Intervention participants who completed the follow-up survey
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PLANTS
Number analyzed (Participants) | 35
score on a scale | 3.93 [3.73 to 4.13]
Statistical Analysis 1: Comparison: PLANTS; Test type: Other — We calculated the mean and 95% confidence interval using a one sample two-sided t-test against the a priori benchmark of success, which was > 3.75; p = 0.074, t-test, 2 sided — Threshold for statistical significance: <0.05; Mean = 3.93, 95% CI 2-sided [3.73 to 4.13]

2. Primary Outcome: Mean Score on the System Usability Scale
Description: At follow-up, participants will complete the ten-question System Usability Scale (SUS) about PLANTS. Each question uses a five-point Likert scale for responses, coded with a value from 1 (Strongly agree) to 5 (Strongly disagree). The odd-numbered question responses will be reverse coded. All items will be summed and that sum will be multiplied by 2.5 to produce the final SUS value (ranging from 0-100). The higher the computed value, the more useable the intervention.
Time Frame: Approximately 4 months after intervention deployment
Population: Intervention participants who completed the follow-up survey
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PLANTS
Number analyzed (Participants) | 35
score on a scale | 75.47 [71.12 to 79.83]
Statistical Analysis 1: Comparison: PLANTS; Test type: Other — We calculated the mean and 95% confidence interval using a one sample two-sided t-test against the a priori benchmark of success, which was > 75; p = 0.827, t-test, 2 sided — Threshold for statistical significance: <0.05; Mean = 75.47, 95% CI 2-sided [71.12 to 79.83]

3. Primary Outcome: Mean Value of Intervention Appropriateness Measure
Description: At follow-up, participants will complete the four-question Intervention Appropriateness Measure (IAM) about PLANTS. Each question uses a five-point Likert scale for responses, coded with a value from 1 (Completely disagree) to 5 (Completely agree) and averaged to produce the mean appropriateness value. The minimum possible mean value is 1 and the maximum mean value is 5. The higher the computed mean value, the more appropriate the intervention.
Time Frame: Approximately 4 months after intervention deployment
Population: Intervention participants who completed the follow-up survey
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PLANTS
Number analyzed (Participants) | 35
score on a scale | 4.01 [3.84 to 4.17]
Statistical Analysis 1: Comparison: PLANTS; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.003, t-test, 2 sided — Threshold for statistical significance: <0.05; Mean = 4.01, 95% CI 2-sided [3.84 to 4.17]

4. Primary Outcome: Mean Value of Feasibility of Intervention Measure
Description: At follow-up, participants will complete the four-question Feasibility of Intervention Measure (FIM) about PLANTS. Each question uses a five-point Likert scale for responses, coded with a value from 1 (Completely disagree) to 5 (Completely agree) and averaged to produce the mean feasibility value. The minimum possible mean value is 1 and the maximum mean value is 5. The higher the computed mean value, the more feasible the intervention.
Time Frame: Approximately 4 months after intervention deployment
Population: Intervention participants who completed the follow-up survey
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PLANTS
Number analyzed (Participants) | 35
score on a scale | 4.01 [3.85 to 4.18]
Statistical Analysis 1: Comparison: PLANTS; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.002, t-test, 2 sided — Threshold for statistical significance: <0.05; Mean = 4.01, 95% CI 2-sided [3.85 to 4.18]

5. Secondary Outcome: Trial Participation Rate
Description: The investigators will divide the number of school staff who consent to participate by the total number of school staff who are invited, then multiply by 100 to get a percentage.
Time Frame: Baseline
Measure: Number (95% Confidence Interval); unit: percentage of total school staff
Groups:
- Overall: All individuals who consented to participate in the study
Arm/Group | Overall
Number analyzed (Participants) | 498
percentage of total school staff | 19.9 [16.5 to 23.7]

6. Secondary Outcome: Trial Retention Rate
Description: The investigators will divide the number of school staff who complete the follow-up survey by the total number of school staff who were enrolled, then multiply by 100 to get a percentage.
Time Frame: At follow-up (approximately 4 months after baseline)
Measure: Number; unit: percentage of consented staff
Arm/Group | PLANTS | EMAILS
Number analyzed (Participants) | 69 | 30
percentage of consented staff | 50.7 | 49.3

7. Secondary Outcome: Intervention Demand
Description: The investigators will divide the number of participants who adhere to the PLANTS intervention by the total number of school staff who were enrolled at schools randomly assigned the PLANTS intervention and multiply by 100 to obtain a percentage. Adherence is a composite variable ranging from 0-100% comprised of: 55% for online module completion (based on the number of completed items divided by the total number of items offered); 45% for Live Zoom Event attendance (where each event is 15%).
Time Frame: At follow-up (approximately 4 months after baseline)
Population: Intent-to-treat intervention population
Measure: Number (95% Confidence Interval); unit: percentage of enrolled staff
Arm/Group | PLANTS
Number analyzed (Participants) | 69
percentage of enrolled staff | 60.80 [49.90 to 71.70]

8. Secondary Outcome: Change in Mean Scores on the Active-Empathic Listening Scale
Description: Participants will complete the eleven-item Active-Empathic Listening Scale at baseline and follow-up. Each item uses a seven-point Likert scale for responses, coded from 1 ("never or almost never true") to 7 ("Always or almost always true"). Mean scores will be calculated for all eleven items at each time point. The minimum possible mean value is 1 and the maximum mean value is 7. Higher values represent greater active-empathic listening. The mean scores from baseline will be subtracted from the mean scores from follow-up to produce the change in mean scores. Higher values represent greater increases in active-empathic listening from baseline to follow-up.
Time Frame: Baseline and follow-up (approximately 4 months after baseline)
Population: Participants who completed the follow-up survey
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PLANTS | EMAILS
Number analyzed (Participants) | 35 | 15
units on a scale | 0.22 [0.03 to 0.42] | 0.01 [-0.36 to 0.38]
Statistical Analysis 1: Comparison: PLANTS; Test type: Other — To test for within-arm statistical significance, we used linear mixed models accounting for within-person clustering using random effects. We reported the beta coefficients and 95% confidence intervals; p = 0.03, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = 0.22, 95% CI 2-sided [0.03 to 0.42]
Statistical Analysis 2: Comparison: EMAILS; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.95, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.36 to 0.38]

9. Secondary Outcome: Change in Mean Scores on Self-efficacy Change Objectives for Providing LGBTQ+ Adolescents With Nurturance, Trustworthiness, and Safety
Description: The investigators have developed items pertaining directly to PLANTS' self-efficacy change objectives. Participants will complete each item using a five-point Likert scale, where 1 represents "not at all certain" and 5 represents "extremely certain." Mean scores will be calculated for all items at each time point. The minimum possible mean value is 1 and the maximum mean value is 5. Higher values represent greater self-efficacy. The mean scores from baseline will be subtracted from the mean scores from follow-up to produce the change in mean scores. Higher values represent greater increases in self-efficacy from baseline to follow-up.
Time Frame: Baseline and follow-up (approximately 4 months after baseline)
Population: Participants who completed the follow-up survey
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PLANTS | EMAILS
Number analyzed (Participants) | 35 | 15
units on a scale
  Self-Efficacy in LGBTQ+ Inclusivity, Awareness, and Advocacy | 0.70 [0.46 to 0.95] | 0.45 [0.10 to 0.80]
  Self-Efficacy in Identity-Affirming Practices | 0.26 [0.11 to 0.41] | 0.13 [0.03 to 0.24]
  Self-Efficacy in Inclusivity in Restrooms and Changing Options | 0.43 [0.18 to 0.68] | 0.44 [0.02 to 0.86]
Statistical Analysis 1: Comparison: PLANTS; Test type: Other — To test for within-arm statistical significance of the change in Self-Efficacy in LGBTQ+ Inclusivity, Awareness, and Advocacy, we used linear mixed models accounting for within-person clustering using random effects. We reported the beta coefficients and 95% confidence intervals; p < 0.001, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = 0.70, 95% CI 2-sided [0.46 to 0.95]
Statistical Analysis 2: Comparison: EMAILS; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.01, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = 0.45, 95% CI 2-sided [0.10 to 0.80]
Statistical Analysis 3: Comparison: PLANTS; Test type: Other — To test for within-arm statistical significance of the change in Self-Efficacy in Identity-Affirming Practices, we used linear mixed models accounting for within-person clustering using random effects. We reported the beta coefficients and 95% confidence intervals; p = 0.001, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = 0.26, 95% CI 2-sided [0.11 to 0.41]
Statistical Analysis 4: Comparison: EMAILS; Test type: Other — [test comment as in outcome 9, analysis 3]; p = 0.01, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = 0.13, 95% CI 2-sided [0.03 to 0.24]
Statistical Analysis 5: Comparison: PLANTS; Test type: Other — To test for within-arm statistical significance of the change in Self-Efficacy in Inclusivity in Restrooms and Changing Options, we used linear mixed models accounting for within-person clustering using random effects. We reported the beta coefficients and 95% confidence intervals; p = 0.001, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = 0.43, 95% CI 2-sided [0.18 to 0.68]
Statistical Analysis 6: Comparison: EMAILS; Test type: Other — [test comment as in outcome 9, analysis 5]; p = 0.04, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = 0.44, 95% CI 2-sided [0.02 to 0.86]

10. Secondary Outcome: Change in Mean Scores on the Teacher Bystander Intervention Model in Traditional Bullying Scale
Description: Participants will complete the 16-item Teacher Bystander Intervention Model in Traditional Bullying scale, which has five subscales. Each response will be coded on a scale of 1 to 5, with 1 representing "strongly disagree" and 5 representing "strongly agree." Mean scores will be calculated for all items at each time point. The minimum possible mean value is 1 and the maximum mean value is 5. Higher values represent greater skills related to bystander intervention in bullying. The mean scores from baseline will be subtracted from the mean scores from follow-up to produce the change in mean scores. Higher values represent greater increases in bystander intervention skills from baseline to follow-up.
Time Frame: Baseline and follow-up (approximately 4 months after baseline)
Population: Participants who completed the follow-up survey
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PLANTS | EMAILS
Number analyzed (Participants) | 35 | 15
units on a scale
  Notice the event | -0.23 [-0.50 to 0.04] | -0.24 [-0.55 to 0.07]
  Interpret the event as an emergency | -0.19 [-0.39 to 0.01] | 0.02 [-0.18 to 0.22]
  Accept responsibility for intervening | -0.15 [-0.30 to 0.01] | 0.07 [-0.14 to 0.28]
  Know how to intervene | 0.33 [0.13 to 0.53] | 0.28 [0.01 to 0.55]
  Implement intervention decisions | -0.06 [-0.19 to 0.07] | -0.03 [-0.16 to 0.10]
Statistical Analysis 1: Comparison: PLANTS; Test type: Other — To test for within-arm statistical significance of the change in Notice the Event, we used linear mixed models accounting for within-person clustering using random effects. We reported the beta coefficients and 95% confidence intervals; p = 0.10, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = -0.23, 95% CI 2-sided [-0.50 to 0.04]
Statistical Analysis 2: Comparison: EMAILS; Test type: Other — [test comment as in outcome 10, analysis 1]; p = 0.14, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = -0.24, 95% CI 2-sided [-0.55 to 0.07]
Statistical Analysis 3: Comparison: PLANTS; Test type: Other — To test for within-arm statistical significance of the change in Interpret the Event as an Emergency, we used linear mixed models accounting for within-person clustering using random effects. We reported the beta coefficients and 95% confidence intervals; p = 0.07, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = -0.19, 95% CI 2-sided [-0.39 to 0.01]
Statistical Analysis 4: Comparison: EMAILS; Test type: Other — [test comment as in outcome 10, analysis 3]; p = 0.85, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.18 to 0.22]
Statistical Analysis 5: Comparison: PLANTS; Test type: Other — To test for within-arm statistical significance of the change in Accept Responsibility for Intervening, we used linear mixed models accounting for within-person clustering using random effects. We reported the beta coefficients and 95% confidence intervals; p = 0.06, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.30 to 0.01]
Statistical Analysis 6: Comparison: EMAILS; Test type: Other — [test comment as in outcome 10, analysis 5]; p = 0.51, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.14 to 0.28]
Statistical Analysis 7: Comparison: PLANTS; Test type: Other — To test for within-arm statistical significance of the change in Know How to Intervene, we used linear mixed models accounting for within-person clustering using random effects. We reported the beta coefficients and 95% confidence intervals; p = 0.001, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = 0.33, 95% CI 2-sided [0.13 to 0.53]
Statistical Analysis 8: Comparison: EMAILS; Test type: Other — [test comment as in outcome 10, analysis 7]; p = 0.04, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = 0.28, 95% CI 2-sided [0.01 to 0.55]
Statistical Analysis 9: Comparison: PLANTS; Test type: Other — To test for within-arm statistical significance of the change in Implement Intervention Decisions, we used linear mixed models accounting for within-person clustering using random effects. We reported the beta coefficients and 95% confidence intervals; p = 0.36, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.19 to 0.07]
Statistical Analysis 10: Comparison: EMAILS; Test type: Other — [test comment as in outcome 10, analysis 9]; p = 0.62, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.16 to 0.10]

11. Secondary Outcome: Change in Mean Scores on the Teacher Bystander Intervention Model in Cyberbullying Scale
Description: Participants will complete the 16-item Teacher Bystander Intervention Model in Cyberbullying scale, which has five subscales. Each response will be coded on a scale of 1 to 5, with 1 representing "strongly disagree" and 5 representing "strongly agree." Mean scores will be calculated for all items at each time point. The minimum possible mean value is 1 and the maximum mean value is 5. Higher values represent greater skills related to bystander intervention in cyberbulling. The mean scores from baseline will be subtracted from the mean scores from follow-up to produce the change in mean scores. Higher values represent greater increases in bystander intervention skills from baseline to follow-up.
Time Frame: Baseline and follow-up (approximately 4 months after baseline)
Population: Participants who completed the follow-up survey
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PLANTS | EMAILS
Number analyzed (Participants) | 35 | 15
units on a scale
  Notice the event | -0.15 [-0.32 to 0.02] | -0.21 [-0.55 to 0.12]
  Interpret the event as an emergency | -0.02 [-0.14 to 0.10] | 0.05 [-0.12 to 0.23]
  Accept responsibility for intervening | -0.07 [-0.22 to 0.09] | -0.12 [-0.37 to 0.13]
  Know how to intervene | 0.39 [0.18 to 0.60] | 0.12 [-0.16 to 0.39]
  Implement intervention decisions | -0.01 [-0.22 to 0.20] | 0.14 [-0.16 to 0.44]
Statistical Analysis 1: Comparison: PLANTS; Test type: Other — [test comment as in outcome 10, analysis 1]; p = 0.08, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.32 to 0.02]
Statistical Analysis 2: Comparison: EMAILS; Test type: Other — [test comment as in outcome 10, analysis 1]; p = 0.20, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = -0.21, 95% CI 2-sided [-0.55 to 0.12]
Statistical Analysis 3: Comparison: PLANTS; Test type: Other — [test comment as in outcome 10, analysis 3]; p = 0.74, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.14 to 0.10]
Statistical Analysis 4: Comparison: EMAILS; Test type: Other — [test comment as in outcome 10, analysis 3]; p = 0.55, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.12 to 0.23]
Statistical Analysis 5: Comparison: PLANTS; Test type: Other — [test comment as in outcome 10, analysis 5]; p = 0.40, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.22 to 0.09]
Statistical Analysis 6: Comparison: EMAILS; Test type: Other — [test comment as in outcome 10, analysis 5]; p = 0.36, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.37 to 0.13]
Statistical Analysis 7: Comparison: PLANTS; Test type: Other — [test comment as in outcome 10, analysis 7]; p < 0.001, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = 0.39, 95% CI 2-sided [0.18 to 0.60]
Statistical Analysis 8: Comparison: EMAILS; Test type: Other — [test comment as in outcome 10, analysis 7]; p = 0.41, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.16 to 0.39]
Statistical Analysis 9: Comparison: PLANTS; Test type: Other — [test comment as in outcome 10, analysis 9]; p = 0.92, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.22 to 0.20]
Statistical Analysis 10: Comparison: EMAILS; Test type: Other — [test comment as in outcome 10, analysis 9]; p = 0.37, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = 0.14, 95% CI 2-sided [-0.16 to 0.44]

12. Secondary Outcome: Change in Mean Scores on the Modified Gay Affirmative Practice Scale
Description: The investigators have modified the language of the Gay Affirmative Practice Scale to incorporate school-oriented words instead of therapy-oriented words to measure self-efficacy for school staff working with SGMY. Participants will complete the nine-item scale at baseline and follow-up, with each item using a five-point Likert scale ranging from "strongly disagree" (1) to "strongly agree" (5). Mean scores will be calculated for all items at each time point. The minimum possible mean value is 1 and the maximum mean value is 5. Higher values represent greater self-efficacy. The mean scores from baseline will be subtracted from the mean scores from follow-up to produce the change in mean scores. Higher values represent greater increases in self-efficacy from baseline to follow-up.
Time Frame: Baseline and follow-up (approximately 4 months after baseline)
Population: Participants who completed the follow-up survey
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PLANTS | EMAILS
Number analyzed (Participants) | 35 | 15
units on a scale | 0.44 [0.28 to 0.59] | 0.49 [0.29 to 0.69]
Statistical Analysis 1: Comparison: PLANTS; Test type: Other — [test comment as in outcome 8, analysis 1]; p < 0.001, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = 0.44, 95% CI 2-sided [0.28 to 0.59]
Statistical Analysis 2: Comparison: EMAILS; Test type: Other — [test comment as in outcome 8, analysis 1]; p < 0.001, Mixed Models Analysis — Threshold for statistical significance: <0.05; Mean Difference (Net) = 0.49, 95% CI 2-sided [0.29 to 0.69]

13. Secondary Outcome: Safety Outcomes
Description: Investigators assess myriad safety outcomes including parent backlash, social media backlash, school board backlash, suspension or removal from employment, censorship of LGBTQ+ literature/history/stories or removal of books with LGBTQ+ representation from school libraries, and emotional discomfort with intervention and control conditions at follow-up. Response options include frequency of each event occurrence (none, once, twice, 3-9 times, and 10 or more times). Investigators will report the overall frequency of events, frequency of each type of event, and percentage of school staff reporting any event.
Time Frame: At follow-up (approximately 4 months after baseline)
Measure: Number; unit: events
Arm/Group | PLANTS | EMAILS
Number analyzed (Participants) | 35 | 15
events
  Overall number of events | 6 | 8
  Times contacted by parents/guardians because there was too much LGBTQ+ inclusivity in school | 0 | 1
  Times contacted by people who were upset because you supported LGBTQ+ students | 0 | 0
  Times your school was attacked for supporting LGBTQ+ youth | 0 | 6
  Times your school board got upset or concerned about staff supporting LGBTQ+ youth | 0 | 0
  Times received negative consequences from your employer about supporting LGBTQ+ youth | 0 | 0
  Times LGBTQ+ censorship happened in your school | 0 | 0
  Times uncomfortable while participating in the course | 6 | 1

ADVERSE EVENTS:
Time Frame: From baseline survey to follow-up survey (seven months)
Arm/Group | PLANTS | EMAILS
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/30
Other Adverse Events (participants affected / at risk) | 0/69 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT05897827/Prot_SAP_000.pdf